CLINICAL TRIAL: NCT06254937
Title: The Effect of Reproductive Life Planning Education on University Students' Fertility and Preconceptional Health Knowledge and Attitudes: Randomized Controlled Study
Brief Title: Fertility and Preconceptional Health Knowledge and Attitudes Among University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ebru Cirban Ekrem (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Ebru Cirban Ekrem, Lecturer, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ege University
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Reproductive Health
Keywords: Reproductive Life Plan; University Student; fertility; Preconceptional Health; Information; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This study was designed as a pretest-posttest randomized controlled experimental study. The research will be conducted in a randomized parallel controlled design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enterprise group (Experimental): The research will be conducted as a randomized controlled trial with a pretest-posttest design.
  Intervention Group: Participants in the intervention group will be given group training based on the contents of the booklet created by the researcher in line with the literature. Training will be given to participants face to face for 40 minutes, once a week for five weeks. Each training session will include two topics in Reproductive Life Plan Based Training Booklet.
  Control Group: A pre-test will be applied to the control group. Reproductive Life Plan Based Training Booklet will be given after the final test.
  Post Intervention Phase After the pre-test is applied to the participants in both groups, the data collection form will be applied again 8 weeks later and the post-test phase of the research will be completed. Participants in the control group will be given Reproductive Life Plan Based Training Booklet.
  Interventions: Other: Reproductive Life Plan training
- control group (No Intervention): Control Group: A pre-test will be applied to the control group. After the final test, the Reproductive Life Plan Based Training Booklet will be given.
  Post Intervention Phase Following the application of the pre-test to the participants in both groups, the data collection form will be applied again 8 weeks later and the post-test phase of the research will be completed. Participants in the control group will be given the Reproductive Life Plan Based Training Booklet after the post-test.

INTERVENTIONS:
Other: Reproductive Life Plan training — Reproductive Life Plan trainings; It will be done in the form of group training, which is considered an advantageous health education method in terms of low cost, wide scope and practicality. During the training, after the power point presentation to the initiative group, question-answer, discussion, brainstorming and visualizations will be made with the Pecha Kucha Technique. Presentations prepared in line with the Reproductive Life Plan Training Booklet will be used as training tools. Training will be given to participants face to face for 40 minutes, once a week for five weeks. Each training session will include two topics in booklet.
  Arms: enterprise group

SUMMARY:
Fertility means being fertile, that is, having the ability to reproduce. Fertility awareness means that individuals know and avoid the anatomy and physiology of the reproductive system, the importance of fertility, fertility options and life habits that negatively affect fertility. Reproductive Life Plans (RLP) are personal goals related to individuals' decisions to have children, when and how to make this decision, focusing on their priorities, current situations and goals.RLP prioritizes preconception care so that individuals can achieve their reproductive goals. This study aimed to examine the effect of RLP training on university students' knowledge and attitudes about fertility and preconception health. The research was designed as a pretest-posttest randomized controlled experimental study. The population of the research will consist of 1025 senior undergraduate students studying in five faculties and 17 departments of Bartın University in the fall semester of the 2023-2024 academic year. To determine the number of participants to be included in the research sample, power analysis was performed using the G-Power 3.1.9.7 program. Accordingly, the sample of the study was planned to include a minimum of 160 participants in intervention and control groups, 80 for each group. Firstly, a Preliminary Evaluation Form will be applied to university students to collect the data of the research. Then, students who meet the inclusion criteria will be pre-tested with the Introductory Information Form, Fertility Health Information Scale and Preconceptional Health Information and Attitude Form. After the pre-test is administered, participants will be randomly assigned to intervention and control groups. Participants in the intervention group will be given group training based on the contents of the Reproductive Life Plan Training Booklet (RLPTB) created by the researcher in line with the literature. No intervention will be made to the participants in the control group. After the pre-test is applied to the participants in both groups, the data collection form will be applied again 8 weeks later and the post-test phase of the research will be completed. IBM SPSS 22.0 package program will be used for statistical analysis of the data obtained from the study. The findings will be evaluated at a 5.0% significance level within a 95.0% confidence interval.

DETAILED DESCRIPTION:
Fertility means being fertile, that is, having the ability to reproduce. Fertility awareness means that individuals know and avoid the anatomy and physiology of the reproductive system, the importance of fertility, fertility options and life habits that negatively affect fertility. Since individuals with fertility awareness have a good level of knowledge about fertility, they are also aware that they should plan pregnancy whenever they want and avoid pregnancy whenever they wish. Reproductive life plan (RLP) is the individual's personal goals related to their decision to have children, when and how they will make this decision, focusing on individuals' priorities, current situations and goals. The aim of the RLP is for both women and men to think about their reproductive intentions, find strategies for successful family planning, and protect themselves from unwanted pregnancies and health consequences that may negatively affect reproduction. RLP prioritizes preconception care so that individuals can achieve their reproductive goals. Women who are healthy during the pre-pregnancy period are more likely to have a healthy pregnancy and have healthy children. The Center for Disease Control (CDC) and ACOG recommend that all individuals of reproductive age be encouraged to have an IMP.

Today, irregular nutrition, insufficient physical activity, obesity, smoking, alcohol and substance use show an increasing trend. All these unhealthy lifestyle habits cause negative effects on fertility and pregnancy outcomes. However, in most OECD countries, it is seen that the average age of women at birth increased by 2 to 5 years between 1970 and 2020, and in many OECD countries, the average age of women at first marriage and birth is 30 years and above. Individuals may encounter fertility problems as a result of advancing marriage and childbearing age. With advancing childbearing age, the risk of obstetric and fetal complications, including gestational diabetes, placenta previa, hypertensive diseases of pregnancy, and fetal congenital anomalies, increases in both the mother and the newborn. In addition, postponing the age of becoming a parent is associated with an increase in the incidence of diseases such as obesity, diabetes, hypertension and thyroid, which means that assisted reproductive techniques will be demanded by an increasing number of couples. Considering all this, it seems that the importance given to fertility awareness should increase today.

Preconception Health Care (PHC) is specialized care targeted to women and men of childbearing age before pregnancy to diagnose, treat and counsel medical and social factors that may prevent positive pregnancy outcomes. The aim of PHC is to optimize the health of expectant mothers and fathers, to ensure that they have a healthy pregnancy experience, and to improve the health conditions of the future baby. PHC also contributes to reducing unwanted and/or unplanned pregnancy rates and maternal and child deaths by making fertility planning of individuals. Although women are generally targeted for fertility and pregnancy issues worldwide and in our country, most men state that they are not included in lifestyle arrangements specific to the preconception period in order to protect and improve their health and fertility.

In the Healthy and Quality Life target, one of the Sustainable Development Goals, it is emphasized that maternal and newborn health should be improved, mortality rates should be reduced, reproductive health should be improved, the importance of family planning and the incidence of non-communicable diseases should be reduced. Understanding reproduction and productivity is important for all young adults. Health care providers have a responsibility to educate people about having children and provide unbiased information and reproductive care. Despite this, when the data of the World Health Organization (WHO) on reproductive health are examined, every year, almost half of all pregnancies are unwanted, 6 out of 10 unwanted pregnancies and 3 out of 10 pregnancies end in induced miscarriage, and almost half of all abortions ( 45%) are seen to be carried out in unsafe ways. This situation negatively affects maternal and neonatal mortality and morbidity. In line with these data, it is seen that most pregnancies worldwide result in unwanted pregnancies, miscarriages and abortions, and it is thought that both women and men have difficulties in the decision to become parents. It is clear that individuals need fertility awareness, preconception care and reproductive life plan services to reduce adverse pregnancy outcomes. In the 11th Development Plan, it is stated that importance should be given to protective and preventive health services that will encourage a healthy lifestyle.

University students, considering their age and developmental characteristics; Since they have gained their autonomy and are in the fertile age, they are faced with a choice between reproductive responsibility and the career development process, where sexual life usually begins. Therefore, college students are a highly vulnerable group to experience adverse reproductive health outcomes.

Purpose of the research: This study aimed to examine the effect of TIP training on university students' fertility and preconceptional health knowledge and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Between May 2023 and October 2024, at Bartın University, Department of Art History, Department of History, Department of Turkish Language and Literature, Department of Contemporary Turkish Dialects and Literatures, Department of Computer Technology and Information Systems and Department of Mathematics at the Faculty of Science. , Department of Computer Engineering of the Faculty of Engineering, Architecture and Design, Department of Electrical and Electronics Engineering, Department of Mechanical Engineering, Department of Landscape Architecture and Department of Civil Engineering, Department of Political Science and Public Administration of the Faculty of Economics and Administrative Sciences, Department of International Trade and Logistics , senior undergraduate students studying in the Department of Economics, Department of Business Administration and Department of Management Information Systems and the Department of Islamic Sciences of the Faculty of Islamic Sciences.
* Female students between the ages of 20-35
* Male students between the ages of 20-40
* Single
* Having no children
* Can communicate in Turkish
* Without visual, hearing or mental disabilities
* Those who volunteer to participate in the research will be included.

Exclusion Criteria:

* Those who are pregnant
* Those who work in the field of health or are taking health-related courses
* Department of Art History, History, Department of Turkish Language and Literature, Department of Contemporary Turkish Dialects and Literatures in the Faculty of Letters of the University, Department of Computer Technology and Information Systems and Department of Mathematics in the Faculty of Science, Computer Engineering Department of the Faculty of Engineering, Architecture and Design. Department of Engineering, Department of Electrical and Electronics Engineering, Department of Mechanical Engineering, Department of Landscape Architecture and Department of Civil Engineering, Department of Political Science and Public Administration of the Faculty of Economics and Administrative Sciences, Department of International Trade and Logistics, Department of Economics, Department of Business Administration and Management Information Systems Those studying in departments other than the Department of Islamic Sciences and the Department of Islamic Sciences of the Faculty of Islamic Sciences will be excluded from the scope of the research.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
There is a difference in Fertility Information Score between the intervention and control groups. | 9 weeks
  There is a difference in Fertility Information Score between the intervention and control groups.
There is a difference in Fertility Attitude Score between the intervention and control groups. | 9 weeks
  There is a difference in Fertility Attitude Score between the intervention and control groups.
There is a difference in Preconceptional Health Knowledge Score between the intervention and control groups. | 9 weeks
  There is a difference in Preconceptional Health Knowledge Score between the intervention and control groups.
There is a difference in Preconceptional Health Attitude Score between the intervention and control groups. | 9 weeks
  There is a difference in Preconceptional Health Attitude Score between the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Cirban Ekrem, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the research will be turned into a doctoral thesis. No personal data of the participants will be shared with anyone.